CLINICAL TRIAL: NCT03015896
Title: A Phase I/II Study of the PD-1 Antibody Nivolumab in Combination With Lenalidomide in Relapsed/Refractory Non-Hodgkin's Lymphoma (NHL) and Hodgkin's Disease (HD)
Brief Title: Nivolumab and Lenalidomide in Treating Patients With Relapsed or Refractory Non-Hodgkin or Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Bond, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, David Bond, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-16167; NCI-2016-01966 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-01-03; First posted 2017-01-10 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Grade 3a Follicular Lymphoma; Recurrent Burkitt Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Waldenstrom Macroglobulinemia; Refractory Burkitt Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Lymphoplasmacytic Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Lenalidomide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lenalidomide, nivolumab) (Experimental): Patients receive lenalidomide PO on days 1-21 and nivolumab IV over 60 minutes on days 1 and 15 of courses 1-4 and on day 1 of courses 5-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This I/II trial studies the side effects and best dose of lenalidomide when given together with nivolumab and to see how well they work in treating patients with non-Hodgkin or Hodgkin lymphoma that has come back and does not respond to treatment. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab and lenalidomide may work better in treating patients with non-Hodgkin or Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of lenalidomide and nivolumab in patients with relapsed/refractory non-Hodgkin lymphoma (NHL). (Phase I) II. To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of the combination of lenalidomide and nivolumab in patients with relapsed/refractory NHL. (Phase I) III. To evaluate the feasibility and toxicities of the combination of lenalidomide and nivolumab in patients with relapsed/refractory Hodgkin's disease (HD). (Phase IB) IV. To evaluate the efficacy of the combination of lenalidomide and nivolumab in terms of overall response rate in patients with relapsed/refractory follicular lymphoma (FL) and diffuse large B-cell lymphoma (DLBCL). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the combination of lenalidomide and nivolumab in patients with relapsed/refractory NHL in terms of overall response rate (ORR), duration of response (DOR), progression-free survival (PFS) and overall survival (OS). (Phase I) II. To evaluate the efficacy of the combination of lenalidomide and nivolumab in patients with relapsed/refractory HD in terms of complete response rate (CR). (Phase IB) III. To evaluate the efficacy of the combination of lenalidomide and nivolumab in patients with relapsed/refractory HD in terms of duration of response (DOR), progression-free survival (PFS) and overall survival (OS). (Phase IB) IV. To evaluate the efficacy of the combination of lenalidomide and nivolumab in patients with relapsed/refractory FL and DLBCL in terms of duration of response (DOR), progression-free survival (PFS) and overall survival (OS). (Phase II)

TERTIARY OBJECTIVES:

I. To explore the relationship between prognostic parameters including ki-67 staining, PD-1 staining and cell of origin (activated B-cell or ABC versus germinal center B-cell or GCB) with ORR to the combination of lenalidomide and nivolumab in patients with relapsed/refractory NHL. (Phase I) II. To evaluate and monitor effects on B-, T-, and natural killer (NK)-cell function with the combination of lenalidomide and nivolumab in patients with relapsed/refractory NHL. (Phase I) III. To explore the relationship between prognostic parameters including ki-67 staining, PD-1 staining and cell of origin (activated B-cell or ABC versus germinal center B-cell or GCB) with ORR to the combination of lenalidomide and nivolumab in patients with relapsed/refractory FL and DLBCL. (Phase II) IV. To evaluate and monitor effects on B-, T-, and NK-cell function with the combination of lenalidomide and nivolumab in patients with relapsed/refractory FL and DLBCL. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Patients receive lenalidomide orally (PO) on days 1-21 and nivolumab intravenously (IV) over 60 minutes on days 1 and 15 of courses 1-4 and on day 1 of courses 5-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Histologically confirmed B-cell NHL with any of the following subtypes: DLBCL, mantle cell lymphoma (MCL), FL, marginal zone lymphoma (MZL) and lymphoplasmacytic lymphoma/Waldenstrom's macroglobulinemia (LL/WM), Burkitt's lymphoma (BL); patients with histological transformation to DLBCL from indolent lymphoma, primary mediastinal lymphoma and grey zone lymphoma are eligible
* PHASE I: Histologically confirmed classical or lymphocyte predominant Hodgkin's disease that is relapsed or refractory after at least one prior chemotherapy
* PHASE I: Patients must have received at least one prior therapy; prior autologous stem cell transplant is permitted; patients with DLBCL who have not had prior high-dose therapy (HDT)/autologous stem cell transplant (ASCT) must be ineligible for transplant; prior lenalidomide is not permitted if patients have progressed on therapy
* PHASE IB DOSE EXPANSION: Histologically confirmed classical or lymphocyte predominant Hodgkin's disease
* PHASE IB DOSE EXPANSION: Patients must have received at least one prior therapy; prior autologous stem cell transplant is permitted; patients who have not had prior HDT/ASCT must be ineligible for transplant; prior lenalidomide is not permitted if patients have progressed on therapy
* PHASE II: Histologically confirmed B-cell NHL:

  * Cohort 1: with only de novo DLBCL or transformed indolent Non-Hodgkin's lymphoma (excludes Richter's syndrome).
  * Cohort 2: with only FL of grade 1, 2 or 3a
* PHASE II: Patients must have received at least one prior therapy (in patients with transformed DLBCL must have received at least one prior therapy; prior autologous stem cell transplant is permitted; patients with DLBCL who have not had prior HDT/ASCT must be ineligible for transplant; prior lenalidomide is not permitted if patients have progressed on therapy
* Be willing and able to provide written informed consent/assent for the trial
* Have evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000 /mcL in the absence of transfusion support within 7 days of determining eligibility
* Hemoglobin >= 8 g/dL
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 40 mL/min creatinine clearance
* Serum total bilirubin =< 1.5 X ULN OR except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 X ULN
* Female subject of childbearing potential should have a negative urine or serum pregnancy at screening and within 24 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects should agree to ongoing pregnancy testing during the course of the study and after the end of study therapy; female subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy; males must refrain from donating sperm during study participation and for 120 days after the last dose of study medication
* Willing and able to receive adequate prophylaxis and/or therapy for thromboembolic events
* Be willing and able to understand and give written informed consent and comply with all study related procedures

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; subjects may use topical or inhaled corticosteroids or low-dose steroids (=< 20 mg of prednisone or equivalent per day) as therapy for comorbid conditions; during study participation, subjects may receive systemic or enteric corticosteroids as needed for treatment-emergent comorbid conditions
* Has a known history of active TB (bacillus tuberculosis)
* Hypersensitivity to nivolumab or lenalidomide or any of their excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy; patients must be 4 weeks out from major procedures
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) lymphoma
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; conditions expected to not recur in the absence of an external trigger
* Has an active infection requiring intravenous systemic therapy
* Is unable to swallow capsules or malabsorption syndrome, disease or condition significantly affecting gastrointestinal function
* Clinically significant cardiovascular disease with uncontrolled arrhythmia, New York Association class 3 or 4 congestive heart failure, history of myocardial infarction within 6 months, or prolonged corrected QT (QTc) > 500 msec
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has progressed on prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has progressed on prior therapy with lenalidomide
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has a history of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia or are at a high risk for a thromboembolic event in the opinion of the investigator and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period
* Has a history of prior allogeneic hematopoietic cell transplant with a history of prior Graft Versus Host Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2026-08-09 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events summarized by NCI CTCAE version 4 | Up to 5 years
  Will be assessed and tabulated across all patients who received any treatment with a focus on severe (grade 3+) adverse events and toxicities (ie those deemed at least possibly related to study treatment). Will also assess tolerability of the regimens through assessing the number of patients who required dose modifications and/or dose delays. Will capture the proportion of patients who go off treatment due to adverse events or those who refuse to continue treated for lesser toxicities.
Maximum tolerated dose (MTD) defined as the dose level at which no more than one of 6 patients experiences a dose-limiting toxicity summarized by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | Up to 28 days
  Will be assessed and tabulated across all patients who received any treatment with a focus on severe (grade 3+) adverse events and toxicities (ie those deemed at least possibly related to study treatment). Will also assess tolerability of the regimens through assessing the number of patients who required dose modifications and/or dose delays. Will capture the proportion of patients who go off treatment due to adverse events or those who refuse to continue treated for lesser toxicities.

SECONDARY OUTCOMES:
Complete response rate (CR) in patients | Up to 5 years
  Complete response rate (CR) in patients with relapsed/refractory HD receiving the combination of lenalidomide and nivolumab
Overall Response Rate (ORR) | Up to 5 years
  Overall Response Rate in patients with relapsed/refractory HD receiving the combination of lenalidomide and nivolumab
Overall Survival (OS) | From study entry to the time of death due to any cause, assessed up to 5 years
  Will be evaluated for each of the cohorts and graphically summarized using the methods of Kaplan and Meier.
Progression free survival (PFS) | From study entry to the time of progression and/or death, assessed up to 5 years
  Will be evaluated for each of the cohorts and graphically summarized using the methods of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: David Bond, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu